CLINICAL TRIAL: NCT02109328
Title: A Phase 2 Study of the Aurora Kinase A Inhibitor Alisertib (MLN8237) in Patients With Relapsed or Refractory Transitional-cell Carcinoma of the Bladder and Urothelial Tract
Brief Title: Alisertib in Chemotherapy-pretreated Urothelial Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Fondazione IRCCS Istituto Nazionale dei Tumori, Milano (Other)
Responsible Party: Principal Investigator, Andrea Necchi, Dr., Fondazione IRCCS Istituto Nazionale dei Tumori, Milano
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: UC-Aurora_INT01; 2014-000557-36 (EudraCT Number)
Record Dates: First submitted 2014-04-03; First posted 2014-04-09 (Estimated); Last update posted 2019-04-11 (Actual); Status verified 2019-04

CONDITIONS: Bladder Cancer; Transitional Cell Carcinoma
Keywords: Bladder cancer; Urothelial cancer; Alisertib; Phase 2; Advanced disease
MeSH Terms: conditions — Urinary Bladder Neoplasms; Carcinoma, Transitional Cell | interventions — MLN 8237; Paclitaxel

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- Alisertib + Paclitaxel (Experimental): After the first single arm phase with Alisertib monotherapy (20 patients, primary endpoint: response-rate), 110 patients will be randomized 1:1 in the second part of the trial.
  Interventions: Drug: Alisertib; Drug: Paclitaxel
- Paclitaxel + Placebo (Placebo Comparator): Weekly paclitaxel + oral Placebo
  Interventions: Drug: Paclitaxel; Drug: Placebo

INTERVENTIONS:
Drug: Alisertib — SINGLE-ARM, SINGLE-DRUG PHASE: Alisertib will be given PO in a dosage of 50 mg BID for 7 Days (Days 1-7) of each 21 day treatment cycle.
  In the randomized phase, Experimental arm will consist of the following drugs:
  Alisertib will be given PO in a dosage of 40 mg twice daily on days 1-3, 8-10 and 15-17 of a 28 day cycle.
  Paclitaxel: 60 mg/m2 over 60 minutes on Days 1, 8, and 15 in a 28-day cycle.
  Other Names: MLN8237
  Arms: Alisertib + Paclitaxel
Drug: Paclitaxel — Placebo will be given PO. Paclitaxel will be infused at the dose of 80 mg/m2 IV over a period of 60 minutes on Days 1, 8, and 15 in a 28-day cycle.
  Other Names: Taxol
Drug: Placebo — Placebo oral tablets
  Arms: Paclitaxel + Placebo

SUMMARY:
Background:

Progress in developing new effective therapies in advanced and relapsing urothelial cancer has been stagnant in the last few decades and a paradigm shift is desperately needed. Aurora kinase-A overexpression has been previously described in bladder cancer and spindle checkpoint dysregulation is a common feature of human urothelial carcinoma (UC).

Alisertib (Millennium Inc.) is an orally available, selective small molecule inhibitor of Aurora A kinase. Single agent and combination treatment of MLN8237 with either paclitaxel (TXL) or gemcitabine synergistically reduced UC cell viability compared with either drug alone. Hence, sequential application of MLN8237 and TXL warrants clinical investigation. Phase 1 trials of both single agent and the combination with TXL defined the recommended doses for phase 2 trials.

Methods:

A multistep approach will be adopted for this Phase 2 trial. A single-group run-in phase will be conducted first with Alisertib 50 mg orally BID for 7 days, followed by 14d rest until disease progression. In case of activity, a confirmatory randomized (1:1) trial of weekly TXL plus either Alisertib or Placebo will follow, incorporating efficacy and futility boundaries for early stopping. In a single-blind design, TXL will be given on days 1,8,15 q4wks at the dose of 60 mg/m2 with alisertib and 80 mg/m2 with placebo. Alisertib dose will be 40 mg BID days 1-3, 8-10 and 15-17, q4wks.

In the single-arm phase, primary endpoint (EP) will be Response Evaluation Criteria in Solid Tumors (RECIST) 1.1 response-rate. 20 pts will be accrued, ≥3 responses will be required (10% type I and 20% type II error constraints). An accrual of 110 pts is foreseen in the randomized phase. Primary EP: progression-free survival (PFS), assuming an improvement in PFS from a median of 2.5 months (H0) to a median of 4.5 months (H1) (44% hazard rate reduction, 10% drop out rate).

Eligibility will include diagnosis of metastatic UC and failure of 1-2 CT regimens (single-arm) or 1 prior CT only (randomized phase). A relapse within 6 months of a peri-operative CT will be counted as 1 line. Computed tomography and PET will be done every 2 cycles (2 months). Additional pharmacodynamic and translational analyses are planned on pre- post- blood and tissue samples.

DETAILED DESCRIPTION:
Phase 2 trial. A single-group run-in phase will be conducted first with Alisertib 50 mg orally BID for 7 days, followed by 14d rest until disease progression.

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed diagnosis of transitional cell tumors of the bladder or the urothelium.
* Locally advanced (T3b,N0; every T,N+) or metastatic disease.
* Failure of max.2 chemotherapy regimens for metastatic disease (at least 1 including a platinum compound).
* Neoadjuvant/adjuvant therapy considered if relapse occurred within 6 months of the last cycle of chemotherapy.

Exclusion Criteria:

* Failure to meet the eligibility requirements.
* Serious medical or psychiatric illness likely to interfere with participation in this clinical study.
* Major co-morbidities as specified in the protocol.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 22 (Actual)
Dates: Start 2014-08-28 (Actual); Primary Completion 2015-07-02 (Actual); Study Completion 2016-10-12 (Actual)

PRIMARY OUTCOMES:
Response rate | 2 months
  Single-arm pilot phase:
  In this phase we will accrue 20 patients, that will be assessed for overall response to treatment (as per RECIST v1.1) as the primary study end point.
Progression-free survival | 2 months
  Randomized Phase:
  Progression free survival will be the primary endpoint. It is foreseen in this phase an accrual of 110 patients, equally balanced in the two arms, in about 36 months and an overall study duration of 40 months, over which we expect to observe 101 disease progressions or deaths. This is the number of events necessary to yield 90% power of a one sided logrank test at the 5% significance level in case of an improvement in PFS from a median of 2.5 months (H0) to a median of 4.5 months (H1), corresponding to a 44% hazard rate reduction in the experimental arm compared to control.

SECONDARY OUTCOMES:
To evaluate the safety and tolerability of Alisertib in a population of chemotherapy pretreated patients with UC. | 2 months
  Incidence and nature of adverse events graded according to the Common Toxicity Criteria for Adverse Effects (CTCAE) version 4.03.

OTHER OUTCOMES:
Translational outcomes | 2 months
  Correlation with tissue and circulating biomarkers with the clinical outcome.

CONTACTS AND LOCATIONS:
Overall Officials: Andrea Necchi, MD, Principal Investigator — Fondazione IRCCS Istituto Nazionale dei Tumori, Milano
Locations (1):
- Fondazione IRCCS Istituto Nazionale dei Tumori, Milan, Mi, Italy

REFERENCES:
- [Derived] Necchi A, Pintarelli G, Raggi D, Giannatempo P, Colombo F. Association of an aurora kinase a (AURKA) gene polymorphism with progression-free survival in patients with advanced urothelial carcinoma treated with the selective aurora kinase a inhibitor alisertib. Invest New Drugs. 2017 Aug;35(4):524-528. doi: 10.1007/s10637-017-0440-5. Epub 2017 Feb 3. PMID 28155045
- [Derived] Necchi A, Lo Vullo S, Mariani L, Raggi D, Giannatempo P, Calareso G, Togliardi E, Crippa F, Di Genova N, Perrone F, Colecchia M, Paolini B, Pelosi G, Nicolai N, Procopio G, Salvioni R, De Braud FG. An open-label, single-arm, phase 2 study of the Aurora kinase A inhibitor alisertib in patients with advanced urothelial cancer. Invest New Drugs. 2016 Apr;34(2):236-42. doi: 10.1007/s10637-016-0328-9. Epub 2016 Feb 12. PMID 26873642